CLINICAL TRIAL: NCT00905840
Title: A Randomized, Controlled, Double Blind, Clinical Trial to Treat Patients With Edentulous Mandibles With Two Straumann 3.3mm Ø Bone Level Implants by Comparing Two Different Implant Alloys in Split Mouth Design.
Brief Title: A Study to Treat Patients With Edentulous Mandibles With Two Straumann 3.3mm Diameter Bone Level Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR 04/07
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Jaw, Edentulous
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titanium Zircon implant (Active Comparator): Intervention: each subject will receive two Straumann bone level implants, one implant is fabricated with Titanium Zircon and the other is a grade IV Titanium implant. Both implants will be randomly placed in the interforaminal region of the edentulous mandible, one on the right half and the other in the left part. Both implants will be treated the same way.
  Interventions: Device: Titanium Grade IV implant
- Titanium Grade IV implant (Placebo Comparator): Intervention: each subject will receive two Straumann bone level implants, one implant is fabricated with Titanium Zircon and the other is a grade IV Titanium implant. Both implants will be randomly placed in the interforaminal region of the edentulous mandible, one on the right half and the other in the left part. Both implants will be treated the same way.
  Interventions: Device: Titanium Zircon implant

INTERVENTIONS:
Device: Titanium Zircon implant — The implant surgery is performed under local anesthesia following standard surgical techniques. The surgeon will be supported by one or two assistants.
  The bone will be excavated and prepared for the placement of the implant. After the implant was placed by using a hand ratched or motor drive device, a healing abutment will be inserted to ensure a transmucosal healing.
  Arms: Titanium Grade IV implant
Device: Titanium Grade IV implant — The implant surgery is performed under local anesthesia following standard surgical techniques. The surgeon will be supported by one or two assistants.
  The bone will be excavated and prepared for the placement of the implant. After the implant was placed by using a hand ratched or motor drive device, a healing abutment will be inserted to ensure a transmucosal healing.
  Arms: Titanium Zircon implant

SUMMARY:
The purpose of this study is to assess the change of crestal bone level at the Titanium Zirconium (TiZr) compared to Titanium (grade IV) implant between surgery and 6, 12, 24, and 36 month post surgery.

DETAILED DESCRIPTION:
This is a clinical trial to compare crestal bone level changes, soft tissue parameters, implant success and survival between small diameter implants in edentulous mandibles restored with removable overdentures.

An initial patient evaluation will be conducted to determine wether a patient meets the study inclusion and exclusion criteria.

The edentulous subjects will undergo surgery for placement of two dental implants, the test and control implant. The implants will be placed in the intraforaminal region.

A gingival former will be inserted in the implant after implant placement to ensures a transmucosal healing. After 6 to 8 weeks the healing abutments will be retrieved and the locator abutments will be connected to the implant.

The removable prosthesis will be prepared and connected to the implants two weeks later.

The study will be blinded until 12 month post surgery and completed with an unblinded follow up period up to 3 years.

Straumann will deliver the randomization envelopes to the sites which had been created by an independent Clinical Research Organization (CRO). The randomization envelopes are marked with a sequential number. The master randomization list will be kept at Straumann.

The success and survival of the implants, soft tissue conditions, success of the prosthesis part and product safety will be assessed after 6, 12, 24, and 36 month after surgery.

Source data verification will be performed by qualified study monitors to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources.

Data will be recorded on standardized Case Report Forms for all study subjects from whom informed consent is obtained. The investigator will be responsible for the accuracy of the data entered on the Case Report Forms. All source documents pertaining to this study will be maintained by the investigator and made available for inspection by authorized persons.

Sample size calculations are proceeded for a given range of clinical relevant differences between test and control implant and a given range of standard deviations with the two sided paired t-test under a significance level of 0.05 and with a power of 80 percent.

To be robust against deviations from the assumption of normality and to take into account possible dropouts it is good clinical practice to increase the calculated sample size by about 10 to 20 percent.

To detect a clinical relevant difference down to 0.1 with a standard deviation of 0.3, one needs 73 plus 15 (88) patients for the study.

Management of dropouts and missing data will depend on their frequency and the particular outcome measure. Any such adjustments will be described completely. All data will be included in the analysis. If outliers are determined to exist, an additional analysis excluding such outliers may be performed and the rationale for such exclusion will be described completely.

A first data analysis including data up to 12 month after surgery is planned after all patients have completed the respective study period. Inferential statistical analysis at this stage will be restricted to the primary efficacy parameter. The final data analysis will be performed after all patients have completed the study.

Categorical data will be described as contingency tables with frequencies and percentage, whereby the dominator for percentages is defined as the number of patients in the respective analysis set. Continuous data will be summarised by mean, standard deviation, minimum, 1st quartile, median, 3rd quartile and maximum. Also the number of missing and nonmissing values will be given.

Tables will be presented by device type and or total, as appropriate. Preabutment connection values will serve as baseline values. Hypothesis tests will be carried out at a two sided significance level of 5 percent, except for the primary efficacy analysis. The confirmatory noninferiority test will be performed at a one sided 2.5 percent significance level.

As usual for secondary, no adjustment os significance level for multiple testing will be performed.

In case of unacceptable deviations from the statistical model assumption, transformations of the data, the use of different distributional models or nonparametric approaches will be considered.

All statistical calculations and analyses will be performed using the Statistical Analysis System (SAS) version 9.1.13 or higher.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have voluntarily signed the informed consent form
* Males and females must be 18 years of age.
* Patients must present with an edentulous mandible at the time of surgery.
* The last tooth or teeth in the mandible must have been extracted or lost more than 8 weeks before the date of first stage surgery.
* The opposing dentition must be edentulous with a denture (implant borne or conventional) or natural or restored teeth
* Adequate bone height of at least 9 mm above vital structures (because the minimal available implant lengths is 8mm) in the intraforaminal region. Available bone width should be in such way that 3.3 mm implants can be placed without the use of concurrent bone augmentation techniques. Harvested bone from the drilling sites may be used to cover minor dehiscence defects.
* Patients must be committed to participate in the study for three years of follow-up examinations

Exclusion Criteria:

* Medical conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* Patients with sever hemophilia
* History of head and neck radiation or chemotherapy
* Patients with history of renal failure
* The application of bisphosphonate medication
* History of uncontrolled endocrine disorders
* Physical handicaps that would interfere with the ability to perform adequate oral hygiene
* Use of any investigational drug or device within the 30-day period immediately prior to implant surgery on study day 0.
* Alcoholism or drug abuse
* Patients with known infection of HIV
* Patients who smoke more than 10 cigarettes per day or cigar equivalents, or who chew tobacco (not greater than 10 cigarette equivalents)
* Fertile females with no adequate method of birth control (contraceptive pill, barrier method, etc.)
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Al-Nawas, PD Dr., Principal Investigator — J. Gutenberg University
Locations (8):
- Catholic University Leuven School of Dentistry, Leuven, Belgium
- Germany (2):
  - J. Gutenberg University, Oral and Maxillofacial Surgery, Mainz
  - Klinikum der Universität Regensburg, Regensburg
- Universitá degli Studi di Milano, Milan, Italy
- Netherlands (2):
  - Academic Center for Dentistry Amsterdam (ACTA), Amsterdam
  - University Medical Center Groningen- UMCG, Groningen
- Switzerland (2):
  - Université de Genève- Section médicine dentaire, Geneva
  - Kantonsspital Luzern, Lucerne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Titan Grade IV Implant and Titan Zircon Implant: Patients with edentulous mandibles received two Straumann bone-level implants, one of Ti Grade IV and one of Titan Zircon in the interforaminal region.
Period: Overall Study
Arm/Group | Titan Grade IV Implant and Titan Zircon Implant
Started | 91
Completed | 75
Not Completed | 16
Not completed — Lost to Follow-up | 11
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Patients with edentulous mandibles
Groups:
- Two Bone Level Implants in Interforaminal Region: All patients received two Straumann bone-level implants, one of Titan Grade IV and one of Titan Zircon alloy. All implants were 3.3 mm in Ø, had a similar macro- and micro-structure, and had the chemically modified SLActive (Sand blasted Large grid Acid-etched) surface.
  The implants were placed in the interforaminal region of the mandible, one implant in each side.
  Implant placement was double-blinded as the implants are visually identical, and the study was unblinded after 12 month for the first analysis.
Arm/Group | Two Bone Level Implants in Interforaminal Region
Number analyzed (Participants) | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 42
Region of Enrollment [Number; unit: participants]
  Belgium | 17
  Netherlands | 12
  Germany | 28
  Italy | 14
  Switzerland | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Crestal Bone Level Between Surgery and 12 Months, to Compare Between the Titan Zircon Implant and the Titan Grade IV Implant.
Description: Panoramic radiographs with standardized setting were taken at the implant surgery and after 12 month. Digital images were analyzed using Image J 1.33 open software and film-based images were digitalized via a video camera, light box and an image analysis program, as described by Braegger (1998; Braegger at al. 2004). All images were analyzed by an independent investigator who was blind to the implant material.
  The implant length was used as a reference measurement, and the implant chamfer 0.2 mm above the implant shoulder was used as the reference line for the bone-level measurement. Bone level was, therefore, defined as the distance from the reference point to the first bone-to-implant contact; mesial and distal bone-level changes in this region were considered as remodeling. Mesial and distal measurements were recorded and the mean of the two values was used.
Time Frame: 12 months
Population: The Intent To Treat (ITT) populaton consisted of all randomized patients who received implants and who underwent at least one efficacy assessment.
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: implants
Groups:
- Titan Grade IV Implant; Titan Zirkon Implant: split-mouth
  Patients with edentulous mandibles received two Straumann bone-level implants, one of Ti Grade IV and one of Ti-Tr, in the interforaminal region. Implants were loaded after 6-8 weeks and removable Locator-retained overdentures were placed within 2 weeks of loading. Modified plaque and sulcus bleeding indices, radiographic bone level, and implant survival and success were evaluated up to 36 month.
Arm/Group | Titan Grade IV Implant | Titan Zirkon Implant
Number analyzed (Participants) | 89 | 89
Number analyzed (implants) | 89 | 89
mm | 0.3 [-0.31 to 0.56] | 0.1 [-0.34 to 0.54]
Statistical Analysis 1: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Null hypothesis: Change of functional bone level at the test implant 12 month after surgery is more than 0.1 lower (inferior) than change of functional crestal bone level at the control implant 12 month after surgery. H-1: Change of functional bone level at the tst implant 12 month after surgery is up to 0.1 lower, equal, or higher (not inferior) than change of functional crestal bone level at the control implant 12 month after surgery; Test type: Non-Inferiority or Equivalence — The analysis of the primary outcome variable, was based on a confirmatory non-inferiority test with a one-sided 97.5% confidence interval. The non-inferiority margin for a clinically relevant difference was set at 0.1 mm. For a sample size of st least 73, a paired t-test with a 0.0025 one-sided significant level was calculated to have 80% power to reject the hypothesis that the test is inferior to the standard; p = 0.025, Student's t-test; Mean Difference (Final Values) = 0.1, 97.5% CI 2-sided [0.1 to 0.3]

2. Secondary Outcome: Success and Survival Rate of Both Study Implants Titanium Grade IV and Titanium Zirconium) According to Definition by Buser et al. 1990
Description: split-mouth design
  Implant success and survival rate according the definition by Buser et al. 1990 are:
  * Absence of persistent subjective complaints, such as pain, foreign body sensation and/or dysaesthesia
  * Absence of a recurrent peri-implant infection with suppuration
  * Absence of mobility
  * Absence of a continuous radiolucency around the implant
  * Possibility for restoration
Time Frame: at 12, 24 and 36 months post surgery
Population: The analysis was determined as Intent To Treat (ITT). The study population consisted of each randomized patient who received the device.
Measure: Number; unit: implants
Units Other Than Participants: implants
Groups:
- Titan Grade IV Implant; Titan Zirkon Implant: split-mouth design
  Patients with edentulous mandibles received two Straumann bone-level implants, one of Ti Grade IV and one of Ti-Tr, in the interforaminal region. Implants were loaded after 6-8 weeks and removable Locator-retained overdentures were placed within 2 weeks of loading. Modified plaque and sulcus bleeding indices, radiographic bone level, and implant survival and success were evaluated up to 36 month.
Arm/Group | Titan Grade IV Implant | Titan Zirkon Implant
Number analyzed (Participants) | 89 | 89
Number analyzed (implants) | 89 | 89
implants
  survival and success rates at 12 month | 84 | 86
  survival and success rates at 24 month | 79 | 80
  survival and success rates at 36 month | 73 | 74
Statistical Analysis 1: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; This analysis is up to 12 month; Test type: Superiority or Other; p = 0.1573, McNemar

3. Secondary Outcome: Soft Tissue and Safety Assessments
Description: Modified Plaque Index (mPI) and modified Sulcus Bleeding Index (mSBI) according to Mombelli at al. (1987). Assessment to be perform at four sites per implant: lingual, buccal, mesial, and distal.
  mPI: 0=no plaque detected, 1=plaque only recognized by running a probe across the smooth marginal surface of the implant, 2=plaque can be seen by the naked eye, 3=abundance of soft matter.
  mSBI: 0=no bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant, 1=isolated bleeding spot visible, 2=blood forms a confluent red line on margin, 3=heavy or profuse bleeding.
  Safety evaluations including recording of all complications, adverse events (AEs), and serious adverse events SAEs). Each AE and SAE will be assessed for severity and its potential relationship to the study device.
Time Frame: after 12, 24, and 36 month
Population: The numbers represent subjects that are classified as Yes. mPI: if all 4 evaluated scores are 0 or 1, the mPI will be classified as No. If at least one score is 2 or 3, mPI will be classified as Yes.
  mSBI: if all evaluated scores are 0 or 1, mSBI will be classified as No. If at least one score is 2 or 3, mSBI will be classified as Yes.
Measure: Number; unit: participants
Arm/Group | Titan Grade IV Implant | Titan Zirkon Implant
Number analyzed (Participants) | 89 | 89
participants
  Plaque Index 12 month | 20 | 19
  Sulcus Beeding Index 12 month | 10 | 9
  Plaque Index 24 month | 16 | 18
  Sulcus Beeding Index 24 month | 7 | 9
  SulcusPlaque Index 36 month | 20 | 19
  Sulcus Beeding Index 36 month | 14 | 13
Statistical Analysis 1: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 0.3617, Wilcoxon (Mann-Whitney) — 12 month data Plaque index
Statistical Analysis 2: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 0.7068, Wilcoxon (Mann-Whitney); 24 month data Plaque index
Statistical Analysis 3: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 0.4312, Wilcoxon (Mann-Whitney); 36 month data Plaque Index
Statistical Analysis 4: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 0.9933, Wilcoxon (Mann-Whitney); 12 month data Sulcus Bleeding Index
Statistical Analysis 5: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 0.3667, Wilcoxon (Mann-Whitney); 24 month data Sulcus Bleeding Index
Statistical Analysis 6: Comparison: Titan Grade IV Implant vs Titan Zirkon Implant; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney); 36 month data Sulcus Bleeding Index

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected 4 weeks after informed consent taken. At visit #2, then at Visit #3; 1-2 weeks after visit #2. 5-6 weeks after visit#3 and 2 weeks after visit #4. Then at 6, 12, 24, and 23 month follow up visits after visit #2.
Groups:
- Two Bone Level Implants in Interforaminal Region: Patients with edentulous mandibles received two Straumann bone-level implants, one of Titan Grade IV and one of Titan Zircon, in the interforaminal region. Implants were loaded after 6-8 weeks and removable Locator-retained overdentures were placed within 2 weeks of loading. Modified plaque and sulcus bleeding indices, radiographic bone level, and implant survival and success were evaluated up to 36 month.
Arm/Group | Two Bone Level Implants in Interforaminal Region
Serious Adverse Events (participants affected / at risk) | 14/91
Other Adverse Events (participants affected / at risk) | 47/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Bone Level Implants in Interforaminal Region (N=91)
New diagnosis breast cancer (Reproductive system and breast disorders) | 1 (2)
Sudden Death (General disorders) | 1 (2) — Reason was not available
Osteomyelitis (Infections and infestations) | 1 (1)
Hypertension (Cardiac disorders) | 1 (2) — Implantation of coronary stent
Vein thrombosis (Vascular disorders) | 1 (1) — Proximal vein thrombosis.
Cervical fracture (Injury, poisoning and procedural complications) | 1 (1) — Patient experienced a severe traumatism on cervical spine.
Myocardial infarction (Cardiac disorders) | 1 (1)
Aneurism (Vascular disorders) | 1 (1) — Abdominal aortic aneurism.
Thyroid neoplasm (Endocrine disorders) | 1 (1) — The thyroid neoplasm resulting in patients death.
Partial knee replacement (Surgical and medical procedures) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) — Patient experienced a life threatening sepsis with pulmonary infection from the precedent cystitis.
Dementia (Nervous system disorders) | 1 (1)
Hip replacement (Surgical and medical procedures) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Two Bone Level Implants in Interforaminal Region (N=91)
Abutment breakage (Surgical and medical procedures) | 1 (1)
Broken arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchopulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Candidiasis (Infections and infestations) | 2 (2)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Chronic pain (General disorders) | 1 (1)
Chronic depression (Psychiatric disorders) | 1 (1)
Costal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Damage of adjacent or opposing dentition (Surgical and medical procedures) | 2 (2)
Denture damage due to accident (Injury, poisoning and procedural complications) | 1 (1)
Fever (General disorders) | 1 (1)
Framework fracture (Surgical and medical procedures) | 9 (9)
Gout (Metabolism and nutrition disorders) | 1 (1)
Granuloma (General disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Infection mycotic (Infections and infestations) | 1 (1)
Infectious colitis (Gastrointestinal disorders) | 1 (1)
Leukoplakia oral (General disorders) | 1 (1)
Loosing of a prosthetic component (Surgical and medical procedures) | 4 (4)
Minor inflammation during the healing process at implant site (Infections and infestations) | 5 (5)
Moderate periimplant infection (Infections and infestations) | 3 (3)
Myositis on leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Opposing framework fracture (Surgical and medical procedures) | 1 (1)
Other minor discomforts due to surgical procedure (Surgical and medical procedures) | 2 (2)
Peridontitis (Infections and infestations) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Prostatitis (Infections and infestations) | 1 (1)
Radiolucency around implant (Musculoskeletal and connective tissue disorders) | 2 (2)
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 2 (2)
Stomatitis (Infections and infestations) | 2 (2)
Tactile horizontal or vertical implant mobility (Musculoskeletal and connective tissue disorders) | 5 (5)
Tooth removal (Surgical and medical procedures) | 3 (3)
Transfer piece fracture (Surgical and medical procedures) | 1 (1)
Worsening diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Wound healing delayed (Infections and infestations) | 1 (1)
Abdominal aortic aneurism (Blood and lymphatic system disorders) | 1 (1)
Osteomyelitis (Injury, poisoning and procedural complications) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Suture removal (Surgical and medical procedures) | 1 (1) — Reason: healing abutment modified.
Surgical uncovering of implant (Surgical and medical procedures) | 1 (1) — Modified procedure.
Spinal operation (Surgical and medical procedures) | 1 (1)
Prosthesis maintenance (Surgical and medical procedures) | 3 (3)
Hypertension (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No